CLINICAL TRIAL: NCT01716689
Title: Phase II Clinical Study of Metronomic Oral Cyclophosphamide in Elderly and/or Pre-treated Patients With Advanced Sarcomas
Brief Title: Clinical Study of Metronomic Oral Cyclophosphamide in Patients With Advanced Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC1201
Record Dates: First submitted 2012-05-13; First posted 2012-10-30 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with advanced sarcoma (Experimental)
  Interventions: Drug: oral cyclophosphamide

INTERVENTIONS:
Drug: oral cyclophosphamide — 50mg daily

SUMMARY:
This is a single arm phase II clinical study to evaluate the efficacy and safety of metronomic oral cyclophosphamide in elderly and/or pre-treated patients with advanced sarcomas.

DETAILED DESCRIPTION:
Eligible patients will receive continuous metronomic oral cyclophosphamide at a dose of 50mg daily. Tumor assessments will be performed at baseline and every 6 weeks thereafter to assess response and disease progression. Toxicity will be monitored throughout treatment. The study's primary end point is defined as clinical benefit rate (CBR) at 12 weeks as a measure of disease control. The study is designed to distinguish a favorable true PFR of 40% from a null rate of 20% [Van Glabbeke et al. EJC 2002]. With a CBR of 40%, metronomic oral cyclophosphamide at this dose and schedule in this patient population will be considered worthy of further evaluation.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate in the study:

1. Participants must have histologically or cytologically confirmed, metastatic and/or unresectable high grade sarcoma for which standard multi-modality curative therapies do not exist or are no longer effective. Patients with low grade sarcoma need to additionally demonstrate disease progression in the last 6 months prior to study entry.
2. Age > 21 years
3. Prior anti-sarcoma chemotherapy

   * Participants who are 21 to 64 years of age at the time of study entry must have received at least one line of established chemotherapy, if such treatment exists; or refused such treatment, which includes either an anthracycline and/or ifosfamide. Patients whose sarcomas do not have known established therapy are eligible for this study without the requirement of a prior therapy.
   * Participants > 65 years of age at the time of study entry are eligible for this study without the requirement for prior treatment
4. ECOG performance status 0-3 (see Annex A)
5. Measurable disease outside of a prior irradiated area as defined by RECIST 1.1 guidelines. A lesion in a previously irradiated area is not eligible for measurable disease unless there is objective evidence of progression of the lesion prior to study enrollment
6. No limit to number of prior chemotherapies or biologics
7. Participants must have normal organ function as defined below:

   * Hemoglobin > 10g/dL
   * Absolute neutrophil count (ANC) > 1500/mm3
   * Platelet count > 75,000/mm3
   * Total bilirubin < 1.5 times institutional upper limits or normal (ULN)
   * AST/ALT < 3 times ULN (< 5 times ULN if hepatic involvement is present)
   * Creatinine < 1.5 times ULN. If creatinine is > 1.5 times ULN, a calculated creatinine clearance time (CCT) should be performed and patient would be eligible for study if the calculated CCT is > 10 mL/min.

   [NB: Glomerular filtration rate (GFR) = [(140 - age) x weight [kg] x 1.22 ] / (serum creatinine [umol/L]. In women, multiply this result by 0.85
8. Resolution, or return to baseline of all clinically significant toxicities related to prior therapies
9. Patients must be suitable for oral drug administration
10. Willingness to use effective means of birth control throughout the duration of clinical study and for at least 3 months after completion of study drug
11. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of study drug administration
12. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.

1. Patients diagnosed with gastrointestinal stromal tumor (GIST)
2. Participants who have had systemic anti-cancer therapy within 3 weeks of study entry (8 weeks for nitrosoureas or mitomycin C)
3. Palliative radiotherapy or major surgery within 3 weeks of study entry
4. Concurrent use of any other anti-cancer therapies or study agents
5. Symptomatic or uncontrolled brain or central nervous system metastases
6. Participants may not be receiving any other concomitant investigational agents
7. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
8. Individuals with a history of a different malignancy, other than cervical cancer in situ, basal cell or squamous cell carcinoma of the skin, are ineligible, except if they have been disease-free for at least 5 years, and are deemed by the investigator to be at low risk for recurrence of that malignancy OR other primary malignancy is neither currently clinically significant nor requiring active intervention.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Clinical benefit as defined by the composite of complete response (CR), partial response (PR) and stable disease (SD) lasting > 12 weeks per RECIST 1.1 as a measure of disease control | 24 months

SECONDARY OUTCOMES:
Assessment of objective response rate (ORR) | 24 months
Assessment of progression free survival | 24 months
Assessment on duration of response to oral metronomic cyclophosphamide in patients who exhibit objective responses | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Quek, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore, Singapore